CLINICAL TRIAL: NCT05320159
Title: Characteristics, Treatment Patterns, and Treatment Satisfaction Among Psoriasis Patients Treated With Cosentyx (Secukinumab)
Brief Title: Treatment Effectiveness Among Psoriasis Patients Treated With Cosentyx (Secukinumab)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457AUS28
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- Overall cohort: Secukinumab: Included all the patients treated with secukinumab
  Interventions: Drug: Secukinumab
- Bio-naive: Included PsO patients initiating treatment with secukinumab. Bio-naïve was defined as no observed treatment (i.e., injection, prescription or patient reported history) with any of the following biologic drugs of interest anytime pre-index: secukinumab, certolizumab, etanercept, adalimumab, infliximab, golimumab, ustekinumab, ixekizumab, brodalumab, abatacept, and guselkumab and risankizumab during all available history
  Interventions: Drug: Secukinumab
- Bio-experienced: Included PsO patients initiating treatment with secukinumab. Patients had pre-index use of one or more of the biologic drugs of interest during all available history
  Interventions: Drug: Secukinumab
- Systemic-naive: Included PsO patients initiating treatment with secukinumab. Systemic-naïve was defined as no observed treatment (i.e., injection, prescription or patient reported history) with any of the biologic treatments or with any of the following systemic (i.e., oral or injectable - no topical forms) drugs of interest pre-index: methotrexate, corticosteroids, acitretin or apremilast.
  Interventions: Drug: Secukinumab
- Systemic-experienced: Included PsO patients initiating treatment with secukinumab. Systemic-experienced patients had pre-index use of one or more of the systemic drugs of interest.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Included all the patients treated with secukinumab
  Other Names: Cosentyx

SUMMARY:
This was a retrospective cohort study utilizing data from Modernizing Medicine Data Services' (MMDS) electronic medical records (EMR)-based dermatology database to evaluate secukinumab patient characteristics, treatment patterns, and outcomes.

DETAILED DESCRIPTION:
This was a retrospective cohort study utilizing data from Modernizing Medicine Data Services' (MMDS) electronic medical records (EMR)-based dermatology database to evaluate secukinumab patient characteristics, treatment patterns, and outcomes. Psoriasis (PsO) patients initiating secukinumab were identified and indexed to the first secukinumab use using the most recent data at study initiation (data period: March 1, 2018 to August 31, 2019) and with a subsequent data refresh (data period: March 1, 2017 - July 31, 2020).

ELIGIBILITY:
Inclusion Criteria:

* ≥1 orders/administrations for secukinumab within the index window (March 1, 2018 to August 31,2019 for the base analysis; March 1, 2018 to January 31, 2020 for the refresh analysis). The date of the first order or administration was be the index date
* Patients in the MMDS database with a diagnosis of PsO on or prior to the 1st secukinumab order/administration
* ≥18 years of age as of the index date
* To ensure capturing continuous patient activities in the EMR dataset, patients must have at least one more visit (any visit regardless of diagnosis) in addition to the index visit within the first 6 months after secukinumab initiation
* Patients must have at least one visit (any visit regardless of diagnosis) within the 12 months pre-index period

Exclusion Criteria:

* Evidence of secukinumab use in the 12-month pre-index period
* Data quality issues (missing age, gender, prescription order information)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients treated with Cosentyx (secukinumab)
Sampling Method: Non-Probability Sample
Enrollment: 17743 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction level at Baseline | Baseline
  Patient reported satisfaction with treatment effectiveness was captured on a 5-point scale - "I believe this treatment is effective in clearing my skin of psoriasis." (1 = strongly agree, 2 = somewhat agree, 3 = Neither agree nor disagree, 4 = Somewhat disagree, 5 = Strongly disagree; n, %) in the EMR data system.
  For this analysis, the responses were classified into three groups:
  1. Satisfied with treatment effectiveness (1 = strongly agree, 2 = somewhat agree)
  2. Dissatisfied with treatment effectiveness ( 4 = Somewhat disagree, 5 = Strongly disagree)
  3. Neither satisfied nor dissatisfied with treatment effectiveness (3 = Neither agree nor disagree)
Treatment satisfaction level at 6 months post-index | 6 months after initiating treatment with secukinumab (The date of the first order or administration was the index date; index period: March 1, 2018 - January 31, 2020)
  Patient reported satisfaction with treatment effectiveness was captured on a 5-point scale - "I believe this treatment is effective in clearing my skin of psoriasis." (1 = strongly agree, 2 = somewhat agree, 3 = Neither agree nor disagree, 4 = Somewhat disagree, 5 = Strongly disagree; n, %) in the EMR data system.
  For this analysis, the responses were classified into three groups:
  1. Satisfied with treatment effectiveness (1 = strongly agree, 2 = somewhat agree)
  2. Dissatisfied with treatment effectiveness ( 4 = Somewhat disagree, 5 = Strongly disagree)
  3. Neither satisfied nor dissatisfied with treatment effectiveness (3 = Neither agree nor disagree)

SECONDARY OUTCOMES:
Age | Baseline (March 1, 2017 - March 1, 2018)
  Age information was reported
Gender | Baseline (March 1, 2017 - March 1, 2018)
  Gender information was reported
Number of patients at various regions | Baseline (March 1, 2017 - March 1, 2018)
  Patient regions: Northeast, Midwest, South, West, Unknown
Number of patients with different race | Baseline (March 1, 2017 - March 1, 2018)
  Race: White, Hispanic, African American, Asian, other/unknown
Weight | Baseline (March 1, 2017 - March 1, 2018)
  Weight of patients was reported
Number of patients at Index year | Study Period: March 1, 2017 - July 31, 2020
  Number of patients at each index year were reported
Number of patients with plaque psoriasis subtype | Baseline (March 1, 2017 - March 1, 2018)
  Plaque psoriasis subtype was categorized as: generalized plaque psoriasis, localized plaque psoriasis, localized scalp psoriasis, inverse psoriasis, palmoplantar psoriasis, guttate psoriasis, nail psoriasis, psoriasis vulgaris, ostraceous psoriasis, or plaque psoriasis with unknown subtype during the 12 month pre-index period (including index date)
Number of patients with Plaque location | Baseline (March 1, 2017 - March 1, 2018)
  Plaque location was categorized as recorded in EMR, including hand, arm, leg, trunk, scalp, head and neck, other/unknown
Comorbidities of interest | Baseline (March 1, 2017 - March 1, 2018)
  Comorbidities of interest during the 12 months pre-index were reported
Physician global assessment (PGA) | Baseline and 6 months post index including index date (The date of the first order or administration was the index date; index period: March 1, 2018 - January 31, 2020)
  PGA is scored on a 6-point scale from 0-5: 0 = clear, 1 = minimal, 2 = mild, 3 =moderate, 4 = marked, and 5 = severe
Total body surface area (TBSA) | Baseline and 6 months post index including index date (The date of the first order or administration was the index date; index period: March 1, 2018 - January 31, 2020)
  Total body surface area (BSA) was expressed as the percentage of body surface involved; BSA values of <3%, 3-10%, and >10% (reported as n, %) will be considered as mild, moderate, or severe, respectively.
Psoriasis-related therapy | 6 months post index including index date (The date of the first order or administration was the index date; index period: March 1, 2018 - January 31, 2020)
  The following categories were included:
  1. Biologics
  2. Methotrexate
  3. Corticosteroids (oral/injection)
  4. Topical therapy
  5. Phototherapy and Psoralen plus ultraviolet A photochemotherapy (PUVA)
  6. NSAID/salicylates
  7. Other systemic plaque psoriasis therapy (Acitretin)
  8. Apremilast (PDE4 inhibitor)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CAIN457AUS28 from the Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17921